CLINICAL TRIAL: NCT00002945
Title: High-Dose Cytarabine and Idarubicin Induction, High Dose Etoposide and Cyclophosphamide Intensification, Autologous Stem Cell Transplantation and Interleukin-2 Immune Modulation in Previously Untreated De Novo and Secondary Adult Myeloid Leukemia
Brief Title: High Dose Chemotherapy, Peripheral Stem Cell Transplantation, and Interleukin-2 in Treating Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065406; RPCI-DS-96-48
Record Dates: First submitted 1999-11-01; First posted 2003-04-16 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Leukemia
Keywords: untreated adult acute myeloid leukemia; adult acute monoblastic leukemia and acute monocytic leukemia (M5); adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute megakaryoblastic leukemia (M7); secondary acute myeloid leukemia; adult acute minimally differentiated myeloid leukemia (M0)
MeSH Terms: conditions — Leukemia; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — aldesleukin; Filgrastim; Cyclophosphamide; Cytarabine; Etoposide; Idarubicin; Melphalan; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: aldesleukin — IV
Biological: filgrastim — IV
Drug: cyclophosphamide — IV
Drug: cytarabine — IV
Drug: etoposide — IV
Drug: idarubicin — IV
Drug: melphalan — IV
Procedure: peripheral blood stem cell transplantation — IV
Radiation: radiation therapy — delivered to the cancer cells

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells. Interleukin-2 may stimulate a person's white blood cells to kill leukemia cells.

PURPOSE: Phase III trial to study the effectiveness of high-dose combination chemotherapy, peripheral stem cell transplantation, and interleukin-2 in treating patients who have acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine relapse free survival of patients with previously untreated de novo or secondary acute myeloid leukemia treated with high dose cytarabine and idarubicin induction, high dose etoposide and cyclophosphamide intensification, filgrastim (G-CSF), melphalan, radiotherapy, autologous peripheral blood stem cell (PBSC) transplantation, and interleukin-2.
* Correlate remission rate and relapse free survival with multidrug resistance phenotype in patients treated with this regimen.
* Determine stem cell content and presence of cells with leukemia specific markers in PBSC harvested following high dose etoposide and cyclophosphamide intensification.
* Correlate NK cell expansion (an increase in both proportion and absolute number) during interleukin-2 therapy following autologous PBSC transplantation with disease free survival.

OUTLINE:

Induction

* Patients receive cytarabine IV over 1 hour every 12 hours for 6 days and idarubicin IV over 30 minutes following third, fifth, and seventh doses of cytarabine. Beginning 12 hours after the last dose of cytarabine, patients receive filgrastim (G-CSF) subcutaneously (SQ) each day until blood counts recover.

Intensification

* Patients receive etoposide IV over 34.3 hours followed 1 hour later by cyclophosphamide IV over 2 hours for 3 days. Beginning 24 hours after the last dose of cyclophosphamide, patients receive G-CSF SQ each day until blood counts recover.

Peripheral blood stem cells (PBSC) are harvested and selected for CD34+ cells. Patients receive melphalan IV over 1 hour on day -4 followed by total body irradiation on days -3, -2, and -1. PBSC are reinfused on day 0.

When blood counts recover, patients receive high dose interleukin-2 SQ on days 1-10 followed by low dose interleukin-2 SQ on days 11-13. Interleukin-2 treatment repeats every 14 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients with immunologic response to 6 courses of interleukin-2 treatment may continue for 6 additional courses.

PROJECTED ACCRUAL: Approximately 100 patients will be accrued for this study over 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven de novo or secondary acute myeloid leukemia with a classification of M0-M2 or M4-M7

  * No classification of M3
  * No promyelocytic leukemia
* Prior medical conditions allowed:

  * Myelodysplastic syndromes
  * Aplastic anemia
  * Paroxysmal nocturnal hemoglobinuria
  * Myeloproliferative disorders except Philadelphia chromosome positive chronic myelogenous leukemia

PATIENT CHARACTERISTICS:

Age:

* Over 25

Performance status:

* Not specified

Life expectancy:

* At least 4 weeks

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 2 times normal
* SGOT no greater than 2 times normal
* Alkaline phosphatase no greater than 2 times normal

Renal:

* Creatinine no greater than 1.5 times normal

Cardiovascular:

* Ejection fraction at least 45%
* No severe cardiovascular disease including myocardial infarction within past 6 months, uncontrolled symptomatic congestive heart failure, angina pectoris, or multifocal cardiac arrhythmias

Other:

* No uncontrolled diabetes mellitus
* No other active malignancy
* No hypersensitivity to E. coli derived drug preparations

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for acute leukemia except hydroxyurea
* Prior chemotherapy allowed for other malignancy or other medical condition

Endocrine therapy:

* Not specified

Radiotherapy:

* Prior radiotherapy allowed for other malignancy or other medical condition

Surgery:

* Not specified

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 1996-12; Primary Completion 2001-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of 4-6 h and 18-24 h, 20% ALA applications on superficial and nodular epidermally-derived lesions using ca633 nm laser irradiation. | 24 hours
  To determine the efficacy of 4-6 h and 18-24 h, 20% ALA applications on superficial and nodular epidermally-derived lesions using ca633 nm laser irradiation.

CONTACTS AND LOCATIONS:
Overall Officials: Meir Wetzler, MD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States